CLINICAL TRIAL: NCT00238797
Title: A Phase II Exploratory, Multicentre, Open-label, Non-comparative Study of ZD1839 (Iressa™) and Radiotherapy in the Treatment of Patients With Glioblastoma Multiforme
Brief Title: A Phase II Exploratory, Multicentre, Open-label, Non-comparative Study of ZD1839 (Iressa) and Radiotherapy in the Treatment of Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0088; D7913L00088 (Other: AZ)
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma multiforme; Brain tumour
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Gefitinib

INTERVENTIONS:
Drug: Gefitinib

SUMMARY:
The purpose of the study is to determine the efficacy of gefitinib (IressaTM) in combination with radiotherapy on patients with glioblastoma multiforme.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* histologically-or cytologically-confirmed glioblastoma multiforme
* age 18 years or older

Exclusion Criteria:

* Have had prior radiation therapy, immunotherapy, gene therapy and/or chemotherapy for the glioblastoma
* co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* known severe hypersensitivity to ZD1839 or any of the excipients of this product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2003-02; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Objective tumour response at 6 months after the end of combination treatment by computerized tomography scan or magnetic resonance imaging of the brain according to Macdonald criteria.

SECONDARY OUTCOMES:
Disease control rate at 6 months after the combination treatment, clinical or radiological progression-free-survival, overall survival and safety of ZD1839 in combination with radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Medical Science Director, MD, Study Director — AstraZeneca
Locations (3):
- Sweden (3):
  - Research Site, Linköping
  - Research Site, Stockholm
  - Research Site, Umeå